CLINICAL TRIAL: NCT02718976
Title: Shamrock - Ultrasound/MR Image Fusion Guided Lumbar Plexus Block
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Bendtsen, Thomas Fichtner, M.D, Ph.D. (Unknown); AP Moeller Foundation (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AUH-TFB-SR-ULMR
Record Dates: First submitted 2016-02-22; First posted 2016-03-24 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-02

CONDITIONS: Hip Fractures; Anesthesia, Local; Pain, Postoperative
Keywords: Hip surgery anesthesia; Perioperative analgesia
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Shamrock guided by US/MR image fusion (Experimental): Use of US/MR image fusion guided Shamrock technique to place lumbar plexus block (20 ml 2% lidocaine with epinephrine added gadoterate meglumine).
  Interventions: Procedure: Ultrasound/MR image fusion guided lumbar plexus block (Shamrock); Drug: Lidocaine-epinephrine added gadoterate meglumine
- Shamrock guided by US (Other): Use of US guided Shamrock technique to place lumbar plexus block (20 ml 2% lidocaine with epinephrine added gadoterate meglumine).
  Interventions: Procedure: Ultrasound guided lumbar plexus block (Shamrock); Drug: Lidocaine-epinephrine added gadoterate meglumine

INTERVENTIONS:
Procedure: Ultrasound/MR image fusion guided lumbar plexus block (Shamrock)
  Arms: Shamrock guided by US/MR image fusion
Procedure: Ultrasound guided lumbar plexus block (Shamrock)
  Arms: Shamrock guided by US
Drug: Lidocaine-epinephrine added gadoterate meglumine — Perineural injection of 20 ml 2% lidocaine with 0.0005% epinephrine added 1 ml of gadoterate meglumine (0.13 ml) and sodium chloride (NaCl, 0.87 ml). The 1 ml of gadoterate meglumine-NaCl is added to the local anesthetic prior to the perineural injection in order to enhance visualization of the local anesthetic on MRI scanning after the intervention.

SUMMARY:
The main objective is to complete a double-blinded randomized controlled crossover trial of lumbar plexus block with the Shamrock technique guided by ultrasound (US)/magnetic resonance imaging (MRI) image fusion vs. the Shamrock technique guided by ultrasound in healthy volunteers.

The investigators will assess block procedure-related parameters, anatomical spread of local anesthetic, and motor and sensory effects.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Body mass index (BMI): 18.5 ≤ BMI ≤30
* Written and oral consent to participate
* Normal healthy person (American Society of Anesthesiology Classification I)

Exclusion Criteria:

* Volunteers not abel to speak or understand Danish
* Volunteers not able to cooperate
* Allergy against the medicines used in the study
* Daily use of analgesics
* Drug abuse - according to the investigator's judgment
* Alcohol consumption greater than the recommendations of the Danish National Board of Health
* Contraindication for MRI scan (including pregnancy)
* Volunteers in whom nerve blocks are impossible due to technical reasons or infection
* Volunteers who are incompetent, eg. surrogate consent is unaccepted

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with a successful block of the femoral and obturator nerves (reduced muscle force compared to baseline assessed with handheld dynamometer), and of the lateral femoral cutaneous nerve (assessed with cold and pinprick test) | Assessed 60 minutes after intervention. Data will be presented 10 months after study completion.
  Block success is defined as the number of volunteers with a successful motor block of the femoral nerve and the obturator nerve, and with a successful sensory block of the lateral femoral cutaneous nerve. Motor block is a proxy marker of sensory block. A participant with a successful motor block has reduced muscle force after block compared to baseline muscle force assessed with handheld dynamometer, and a participant with a successful sensory block has decreased/absent sensation for cold and/or pinprick.

SECONDARY OUTCOMES:
Time for preparation of block procedure (seconds) | Assessed 3 minutes prior to intervention. Data will be presented 10 months after study completion.
  Time for block preparation is defined as the time period from the time point when the volunteer is placed on the block bed to the time point when the pre-ultrasound scanning before intervention is complete.
Time for block procedure (seconds) | Assessed 0 minutes after intervention. Data will be presented 10 months after study completion.
  Time for block procedure is defined as the time period from the time point when the ultrasound probe is placed on the skin after completed preparation to the time point when the block needle is pulled out after injection of local anesthetics (end of intervention).
Electrical nerve stimulation strength (mA) | Assessed 1 minute before injection of injectate. Data will be presented 10 months after study completion.
  Minimal electrical nerve stimulation (mA) required to trigger neuromuscular response and confirm correct placement of block needle prior to injection of local anesthetics.
Electrical nerve stimulation response (quadriceps, sartorius, other muscular, paresthesia, none) | Assessed 1 minute before injection of injectate. Data will be presented 10 months after study completion.
  Type of neuromuscular response on electrical nerve stimulation.
Needle advancements | Assessed 0 minutes after intervention. Data will be presented 10 months after study completion.
  Number of needle advancements during intervention.
Injection site | Assessed 0 minutes after intervention. Data will be presented 10 months after study completion.
Block needle depth | Assessed 0 minutes after intervention. Data will be presented 10 months after study completion.
Discomfort | Assessed 0 minutes after intervention. Data will be presented 10 months after study completion.
  Estimated on numeric rating scale 0-10
Mean arterial pressure change | Mean arterial pressure is measured prior to intervention and 5 min after intervention. Data will be presented 10 months after study completion.
Number of participants with visual confirmed contact between the injectate and the spinal nerves L2-S1, the femoral, the obturator, and the lateral femoral cutaneous nerves, and the lumbosacral trunk assessed on MRI | Assessed on MRI sampled 10-40 minutes after intervention. Data will be presented 10 months after study completion.
Number of participants with visually confirmed epidural spread of the injectate assessed on MRI. | Assessed on MRI sampled 10-40 minutes after intervention. Data will be presented 10 months after study completion.
Number of participants with motor block | Baseline muscle strength is estimated prior to first intervention. Post-block muscle strength is estimated 60 minutes after intervention. Data will be presented 10 months after study completion.
  Muscle strength of the femoral, obturator, superior gluteal, and sciatic nerves are estimated with handheld dynamometer during knee extension, hip adduction, hip abduction, and knee flexion. Motor block is assessed as reduced muscle strength compared to baseline.
Number of participants with sensory block | Estimated 70 minutes after intervention. Data will be presented 10 months after study completion.
  Sensory block is defined as decreased or absent sensation for cold, warmth, touch, and pinprick are assessed for the dermatomes T8-S3 and the lateral femoral cutaneous nerve.
Cost-effectiveness (ICER) | Calculated 1 month after study completion. Data will be presented 10 months after study completion.
  ICER is estimated as the difference in mean marginal cost of the blocks.
Quantitative diffusion weighted MRI reproducibility | Assessed on MRI sampled 40-55 minutes after intervention. Data will be presented 10 months after study completion.
Image evaluation of diffusion weighted MRI reproducibility | Assessed on MRI sampled 40-55 minutes after intervention. Data will be presented 10 months after study completion.

CONTACTS AND LOCATIONS:
Overall Officials: Jennie MC Strid, M.D., Principal Investigator — Department of Anesthesiology and Intensive Care, Aarhus University Offical

IPD SHARING:
Plan to Share IPD: No